CLINICAL TRIAL: NCT03611582
Title: Effect and Safety of Semaglutide 2.4 mg Once-weekly as Adjunct to Intensive Behavioural Therapy in Subjects With Overweight or Obesity
Brief Title: Research Study to Look at How Well Semaglutide is at Lowering Weight When Taken Together With an Intensive Lifestyle Program
Acronym: STEP 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4375; U1111-1200-8199 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide 2.4 mg during 68-week treatment period in addition to intensive behavioural therapy.
  Interventions: Drug: Semaglutide
- Semaglutide placebo (Placebo Comparator): Participants will receive semaglutide placebo during 68-week treatment period in addition to intensive behavioural therapy.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous (s.c., under the skin) injections of semaglutide once weekly at escalating doses (0.25 mg/week, 0.5 mg/week, 1.0 mg/week, 1.7 mg/week, 2.4 mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide
Drug: Placebo (semaglutide) — S.c. injections of placebo once weekly at a similar dose escalation manner as semaglutide (placebo matched to semaglutide 0.25 mg/week, 0.5 mg/week, 1.0 mg/week, 1.7 mg/week, 2.4 mg/week). The dose will be escalated to next level every 4 weeks.
  Arms: Semaglutide placebo

SUMMARY:
This study will look at the change in participant's body weight from the start to the end of the study. This is to compare the effect on body weight in people taking semaglutide (a new medicine) and people taking "dummy" medicine. Together with the medicine, the participant will also be part of an intensive lifestyle program where the participant will have talks with study staff about healthy food choices, what the participant can do to lose weight and be more physically active. The participant will either get semaglutide or "dummy" medicine - which treatment the participant gets is decided by chance. The participant will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. For the first 2 months the participant will be on a low calorie diet. The diet is made up of bars, shakes and 1 low calorie pre-prepared meal for each day. The study will last for about 1.5 years. The participant will have 32 clinic visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age more than or equal to 18 years at the time of signing informed consent
* Body mass index more than or equal to 30 kg/m^2 or more than or equal to 27 kg/m^2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Hemoglobin A1c more than or equal to 48 mmol/mol (6.5%) as measured by the central laboratory at screening
* A self-reported change in body weight more than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (39):
- United States (39):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Evanston, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Endwell, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Rockwall, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Kushner RF, Calanna S, Davies M, Dicker D, Garvey WT, Goldman B, Lingvay I, Thomsen M, Wadden TA, Wharton S, Wilding JPH, Rubino D. Semaglutide 2.4 mg for the Treatment of Obesity: Key Elements of the STEP Trials 1 to 5. Obesity (Silver Spring). 2020 Jun;28(6):1050-1061. doi: 10.1002/oby.22794. PMID 32441473
- [Result] Wadden TA, Bailey TS, Billings LK, Davies M, Frias JP, Koroleva A, Lingvay I, O'Neil PM, Rubino DM, Skovgaard D, Wallenstein SOR, Garvey WT; STEP 3 Investigators. Effect of Subcutaneous Semaglutide vs Placebo as an Adjunct to Intensive Behavioral Therapy on Body Weight in Adults With Overweight or Obesity: The STEP 3 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1403-1413. doi: 10.1001/jama.2021.1831. PMID 33625476
- [Derived] Wadden TA, Brown GK, Egebjerg C, Frenkel O, Goldman B, Kushner RF, McGowan B, Overvad M, Fink-Jensen A. Psychiatric Safety of Semaglutide for Weight Management in People Without Known Major Psychopathology: Post Hoc Analysis of the STEP 1, 2, 3, and 5 Trials. JAMA Intern Med. 2024 Nov 1;184(11):1290-1300. doi: 10.1001/jamainternmed.2024.4346. PMID 39226070
- [Derived] Heerspink HJL, Apperloo E, Davies M, Dicker D, Kandler K, Rosenstock J, Sorrig R, Lawson J, Zeuthen N, Cherney D. Effects of Semaglutide on Albuminuria and Kidney Function in People With Overweight or Obesity With or Without Type 2 Diabetes: Exploratory Analysis From the STEP 1, 2, and 3 Trials. Diabetes Care. 2023 Apr 1;46(4):801-810. doi: 10.2337/dc22-1889. PMID 36801984
- [Derived] Perreault L, Davies M, Frias JP, Laursen PN, Lingvay I, Machineni S, Varbo A, Wilding JPH, Wallenstein SOR, le Roux CW. Changes in Glucose Metabolism and Glycemic Status With Once-Weekly Subcutaneous Semaglutide 2.4 mg Among Participants With Prediabetes in the STEP Program. Diabetes Care. 2022 Oct 1;45(10):2396-2405. doi: 10.2337/dc21-1785. PMID 35724304
- [Derived] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 41 sites in the United States.
Pre-assignment Details: The trial has a 68-week treatment period (16 weeks of dose escalation and 52 weeks of maintenance dose). Participants were randomised in 2:1 ratio either to receive semaglutide 2.4 mg or placebo.
Groups:
- Semaglutide 2.4 mg: Participants were to receive once-weekly subcutaneous (s.c) injection of semaglutide using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL or 3.2 mg/mL in 16 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg and 1.7 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. Treatment was continued on the maintenance dose of 2.4 mg once weekly for an additional 52 weeks until week 68. The treatment was an adjunct to Intensive Behavioural Therapy (IBT), which involves physical activity and dietary intervention with the first 8 weeks of a low-calorie diet (LCD) followed by a strict hypo-caloric diet till the end of treatment.
- Placebo: Participants were to receive once-weekly s.c injection of matching semaglutide placebo using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide placebo 1.0 mg/mL or 3.0 mg/mL or 3.2 mg/mL in 16 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, and 1.7 mg) every fourth week until a maintenance dose of 2.4 mg of semaglutide placebo was reached. Treatment was continued on the maintenance dose of 2.4 mg once weekly for an additional 52 weeks until week 68. The treatment was an adjunct to IBT, which involves physical activity and dietary intervention with the first 8 weeks of LCD followed by a strict hypo-caloric diet till the end of treatment.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 407 | 204
Full Analysis Set (FAS) | 407 | 204
Safety Analysis Set (SAS) | 407 | 204
Completed | 339 | 166
Not Completed | 68 | 38
Not completed — Adverse Event | 26 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Pregnancy | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — At the discretion of the investigator | 1 | 0
Not completed — Safety concern as judged by the investigator | 1 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 18 | 7
Not completed — other | 17 | 16

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 407 | 204 | 611
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (13) | 46 (13) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 180 | 495
  Male | 92 | 24 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 46 | 121
  Not Hispanic or Latino | 332 | 158 | 490
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 80 | 36 | 116
  White | 307 | 158 | 465
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Change in body weight from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from both in-trial and on-treatment periods. In-trial observation period: the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact (week 75). On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomized participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 407 | 204
Percentage
  In-trial observation period: number analyzed (Participants) | 373 | 189
  In-trial observation period | -16.5 (10.1) | -5.8 (7.7)
  On-treatment observation period: number analyzed (Participants) | 334 | 164
  On-treatment observation period | -17.6 (9.6) | -6.1 (7.6)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -10.27, 95% CI 2-sided [-11.97 to -8.57]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority; p < 0.0001, MMRM (mixed model repeated measurement); Treatment difference = -12.67, 95% CI 2-sided [-14.34 to -11.00]

2. Primary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 5%
Description: Number of participants who achieved greater than or equal to (≥) 5% weight loss after 68 weeks is presented. In the reported data, 'Yes' infers the number of participants who have achieved ≥ 5% weight loss, whereas 'No' infers the number of participants who have not achieved ≥ 5% weight loss. The endpoint was evaluated based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75). On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 2 weeks of follow-up. It excludes any period of temporary treatment interruption.
Time Frame: After 68 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 407 | 204
Participants
  In-trial observation period: number analyzed (Participants) | 373 | 189
  In-trial observation period: Yes | 323 | 90
  In-trial observation period: No | 50 | 99
  On-treatment observation period: number analyzed (Participants) | 334 | 164
  On-treatment observation period: Yes | 300 | 82
  On-treatment observation period: No | 34 | 82
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.11, 95% CI 2-sided [4.04 to 9.26]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority; p < 0.0001, MMRM (mixed model repeated measurement); Odds Ratio (OR) = 11.67, 95% CI 2-sided [7.64 to 17.81]

3. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 10%
Description: Number of participants who achieved greater than or equal to (≥) 10% weight loss after 68 weeks is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 10% weight loss whereas 'No' infers number of participants who have not achieved ≥ 10% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: After 68 weeks
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 373 | 189
Participants
  Yes | 281 | 51
  No | 92 | 138

4. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 15%
Description: Number of participants who achieved greater than or equal to (≥) 15% weight loss after 68 weeks is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 15% weight loss whereas 'No' infers number of participants who have not achieved ≥ 15% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: After 68 weeks
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 373 | 189
Participants
  Yes | 208 | 25
  No | 165 | 164

5. Secondary Outcome: Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 20%
Description: Number of participants who achieved greater than or equal to (≥) 20% weight loss after 68 weeks is presented. In the reported data, 'Yes' infers number of participants who have achieved ≥ 20% weight loss whereas 'No' infers number of participants who have not achieved ≥ 20% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: After 68 weeks
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 373 | 189
Participants
  Yes | 133 | 7
  No | 240 | 182

6. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 371 | 189
Centimeter (cm) | -15.2 (10.2) | -6.1 (8.6)

7. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 188
Millimeters of mercury (mmHg) | -6 (14) | -2 (15)

8. Secondary Outcome: Change in Short Form-36 (SF-36) - Physical Functioning Score
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary and mental component summary). The 0-100 scale scores from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively. Change from week 0 in the domain scores and component summary scores were evaluated at week 68. A positive change score indicates an improvement since baseline. These endpoints were evaluated based on the data from in-trial observation period which is the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 407 | 204
Score on a scale
  Change in physical functioning score (SF-36): number analyzed (Participants) | 364 | 181
  Change in physical functioning score (SF-36) | 2.5 (5.7) | 1.7 (5.7)
  Change in SF-36: Role-Physical score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Role-Physical score | 1.6 (6.5) | 1.5 (6.7)
  Change in SF-36: Bodily Pain score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Bodily Pain score | 1.3 (7.1) | 0.6 (8.3)
  Change in SF-36: General Health score: number analyzed (Participants) | 364 | 181
  Change in SF-36: General Health score | 3.4 (6.6) | 1.9 (6.4)
  Change in SF-36: Vitality score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Vitality score | 2.0 (8.2) | 0.9 (7.8)
  Change in SF-36: Social Functioning score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Social Functioning score | 0.1 (6.6) | -1.2 (8.0)
  Change in SF-36: Mental Health score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Mental Health score | -0.5 (6.0) | -1.5 (7.1)
  Change in SF-36: Physical component summary: number analyzed (Participants) | 364 | 181
  Change in SF-36: Physical component summary | 3.2 (6.0) | 2.6 (6.5)
  Change in SF-36: Mental component summary: number analyzed (Participants) | 364 | 181
  Change in SF-36: Mental component summary | -0.9 (6.0) | -2.2 (8.0)
  Change in SF-36: Role-Emotional score: number analyzed (Participants) | 364 | 181
  Change in SF-36: Role-Emotional score | -0.6 (5.6) | -1.5 (7.7)

9. Secondary Outcome: Change in Body Weight (Kg)
Description: Change in body weight from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 373 | 189
Kilogram (kg) | -17.5 (11.4) | -6.2 (8.6)

10. Secondary Outcome: Change in Body Mass Index
Description: Change in body mass index from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/sqm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 373 | 189
Kilogram per square meter (kg/sqm) | -6.2 (4.0) | -2.2 (3.1)

11. Secondary Outcome: Change in HbA1c (%)
Description: Change in glycosylated haemoglobin (HbA1c) from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 369 | 184
Percentage point of HbA1c | -0.5 (0.3) | -0.3 (0.2)

12. Secondary Outcome: Change in HbA1c (mmol/Mol)
Description: Change in HbA1c from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 369 | 184
mmol/mol | -5.8 (3.1) | -3.1 (2.5)

13. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from week 0 to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 355 | 176
milligrams per deciliter (mg/dL) | -7.3 (10.9) | -1.1 (10.6)

14. Secondary Outcome: Change in Fasting Serum Insulin
Description: Change in fasting serum insulin from week 0 to week 68 [measured as milli-international units per milliliter (mIU/mL)] is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 346 | 170
Ratio of fasting serum insulin | 0.68 (67.4) | 0.84 (50.6)

15. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 372 | 188
mmHg | -3 (10) | -1 (10)

16. Secondary Outcome: Change in Total Cholesterol
Description: Change in fasting total cholesterol from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 181
Ratio of fasting total cholesterol | 0.96 (15.0) | 1.01 (12.3)

17. Secondary Outcome: Change in High-density Lipoproteins (HDL)
Description: Change in fasting HDL from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline.The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 181
Ratio of fasting HDL cholesterol | 1.06 (14.6) | 1.05 (15.0)

18. Secondary Outcome: Change in Low-density Lipoproteins (LDL)
Description: Change in fasting LDL from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 181
Ratio of fasting LDL cholesterol | 0.96 (23.2) | 1.01 (18.6)

19. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL)
Description: Change in fasting VLDL from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 181
Ratio of fasting VLDL cholesterol | 0.77 (40.9) | 0.91 (38.6)

20. Secondary Outcome: Change in Free Fatty Acids
Description: Change in fasting free fatty acids from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting free fatty acids
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 346 | 171
Ratio of fasting free fatty acids | 0.86 (69.9) | 1.08 (71.8)

21. Secondary Outcome: Change in Triglycerides
Description: Change in fasting triglycerides from baseline (week 0) to week 68 (measured as mg/dL) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 181
Ratio of fasting triglycerides | 0.77 (41.3) | 0.91 (39.1)

22. Secondary Outcome: Change in High Sensitivity C-reactive Protein
Description: Change in high sensitivity C-reactive protein from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per litre (mg/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 363 | 182
milligrams per litre (mg/L) | 0.40 (108.7) | 0.76 (75.5)

23. Secondary Outcome: Change in Plasminogen Activator Inhibitor-1 Activity
Description: Change in plasminogen activator inhibitor-1 activity from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Arbritary units per milliliter (AU/ml)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 343 | 162
Arbritary units per milliliter (AU/ml) | 0.92 (80.6) | 1.26 (74.2)

24. Secondary Outcome: Participants Who Achieve (Yes/no): Responder Definition Value for SF-36 Physical Functioning Score
Description: The observed number of participants experiencing a meaningful within participant improvement in SF-36 Physical function after 68 weeks was determined based on two thresholds. The threshold of 4.3 is the default generic responder threshold defined in SF-36 manual for a general population. The threshold of 3.7 is specific for overweight or obese population included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on Food and Drug Administration (FDA) recommendations. In the reported data, "Yes" infers number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on the in-trial observation period which is uninterrupted time interval from randomization (week 0) to last trial related subject-site contact (week 75).
Time Frame: After 68 weeks
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 364 | 181
Participants
  Yes (with threshold 4.3) | 86 | 36
  No (with threshold 4.3) | 278 | 145
  Yes (with threshold 3.7) | 133 | 51
  No (with threshold 3.7) | 231 | 130

25. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 8 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 8
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 396 | 197
Percentage | -7.8 (3.1) | -6.0 (3.6)

26. Secondary Outcome: Number of Treatment-emergent Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event that had onset date (or increase in severity) on or after the first day of exposure to treatment. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 75
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 407 | 204
events | 4035 | 1325

27. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. The SAEs occurred from week 0 to week 75 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 75
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 407 | 204
events | 55 | 7

28. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: SAS included all participants who received at least one dose of trial product. Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 334 | 163
beats per minute (bpm) | 3 (11) | 2 (10)

29. Secondary Outcome: Change in Amylase
Description: Change in amylase (measured as U/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 332 | 161
Ratio of amylase | 1.12 (19) | 1.07 (18.1)

30. Secondary Outcome: Change in Lipase
Description: Change in lipase (measured as U/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 332 | 161
Ratio of lipase | 1.31 (52) | 0.94 (39.4)

31. Secondary Outcome: Change in Calcitonin
Description: Change in calcitonin (measured as ng/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 332 | 162
Ratio of calcitonin | 0.93 (40.6) | 0.94 (33.2)

ADVERSE EVENTS:
Time Frame: week 0 to week 75 Results are based on the SAS which included all participants who received at least one dose of semaglutide or placebo.
Description: All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment and no later than the date of last dose + 7 weeks.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/407 | 0/204
Serious Adverse Events (participants affected / at risk) | 37/407 | 6/204
Other Adverse Events (participants affected / at risk) | 379/407 | 177/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=407) | Placebo (N=204)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Neck dissection (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=407) | Placebo (N=204)
Abdominal distension (Gastrointestinal disorders) | 41 (55) | 20 (28)
Abdominal pain (Gastrointestinal disorders) | 53 (75) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 33 (45) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (54) | 19 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 53 (67) | 22 (24)
Constipation (Gastrointestinal disorders) | 150 (210) | 50 (62)
Decreased appetite (Metabolism and nutrition disorders) | 35 (36) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 147 (307) | 45 (62)
Dizziness (Nervous system disorders) | 52 (73) | 11 (14)
Dyspepsia (Gastrointestinal disorders) | 36 (47) | 10 (15)
Eructation (Gastrointestinal disorders) | 36 (52) | 1 (1)
Fatigue (General disorders) | 52 (69) | 15 (19)
Flatulence (Gastrointestinal disorders) | 47 (62) | 23 (24)
Gastroenteritis (Infections and infestations) | 28 (32) | 12 (19)
Gastroenteritis viral (Infections and infestations) | 41 (46) | 13 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 (32) | 4 (4)
Headache (Nervous system disorders) | 78 (123) | 20 (25)
Influenza (Infections and infestations) | 27 (32) | 11 (11)
Nasopharyngitis (Infections and infestations) | 90 (128) | 49 (70)
Nausea (Gastrointestinal disorders) | 237 (511) | 45 (60)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 12 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17) | 13 (14)
Seasonal allergy (Immune system disorders) | 12 (18) | 11 (14)
Sinusitis (Infections and infestations) | 39 (51) | 26 (34)
Upper respiratory tract infection (Infections and infestations) | 85 (115) | 44 (65)
Urinary tract infection (Infections and infestations) | 41 (60) | 10 (11)
Vomiting (Gastrointestinal disorders) | 111 (212) | 22 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03611582/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03611582/SAP_001.pdf